CLINICAL TRIAL: NCT05251610
Title: Does Oral Propranolol Accelerate Labor Induction/Augmentation With Oxytocin in Nulliparous Women in Abakaliki?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darlington-Peter Chibuzor Ugoji (Other)
Responsible Party: Sponsor-Investigator, Darlington-Peter Chibuzor Ugoji, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FETHA/REC/VOL2/2019/277
Record Dates: First submitted 2021-09-22; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Duration of Labor
MeSH Terms: interventions — Propranolol; Oxytocin

STUDY DESIGN:
Intervention Model Description: clinical superiority open-labeled randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROPRANOLOL GROUP (Active Comparator): Participants will receive 20mg of oral propranolol 10 minutes prior to initiation of augmentation or induction of labor with oxytocin
  Interventions: Drug: 20mg oral propranolol and oxytocin
- OXYTOCIN ONLY GROUP (Placebo Comparator): Participants had outright augmentation or induction of labor with oxytocin only
  Interventions: Drug: Oxytocin only

INTERVENTIONS:
Drug: 20mg oral propranolol and oxytocin — Participants will receive 20mg of oral propranolol 10minutes prior to initiation of augmentation or induction of labor with oxytocin
  Arms: PROPRANOLOL GROUP
Drug: Oxytocin only — Participants will have outright augmentation or induction of labor with oxytocin
  Arms: OXYTOCIN ONLY GROUP

SUMMARY:
Labour is usually physiologic, spontaneous and progressive, but occasionally, there may be the need for induction or augmentation of labour especially in nulliparous women, who are at increased risk of dysfunctional labour. Oxytocin traditionally has been used for induction and augmentation of labour however prolonged labour continued to occur with attendant sequelae. Newer agents like propranolol, with minimal to no maternal and fetal adverse effects in labour have been shown to decreases the duration of labour when used in synergy with oxytocin. However, the paucity of information on the use of propranolol in labour.

DETAILED DESCRIPTION:
ABSTRACT Background: Labour is usually physiologic, spontaneous and progressive, but occasionally, there may be the need for induction or augmentation of labour especially in nulliparous women, who are at increased risk of dysfunctional labour. Oxytocin traditionally has been used for induction and augmentation of labour however prolonged labour continued to occur with attendant sequelae. Newer agents like propranolol, with minimal to no maternal and fetal adverse effects in labour have been shown to decreases the duration of labour when used in synergy with oxytocin. However, the paucity of information on the use of propranolol in labour.

Methodology: This research was a superiority open labelled randomized controlled trial that involved only nulliparous women who met the inclusion criteria and gave consent to the study. There was daily recruitment of participants. Randomization was by utilizing computer-generated numbers from a pool of 110 participants divided into A and B. Group A received 20 mg of oral propranolol before initiation of oxytocin titration. Group B received only oxytocin titration. Partograph was used to monitor their labour.

Analysis: Absolute and relative frequencies of categorical variables, mean, range and standard deviation of continuous variables were calculated. Continuous variables were analyzed using students t-test while chi-square (χ2) test was used for categorical variables. A P-value of <0.05 was considered significant.

Keywords: Propranolol, Labour, Induction, Augmentation, Nullipara

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women selected for induction or augmentation of labour
2. Term pregnancy selected for induction or augmentation of labour
3. Normal singleton pregnancies with cephalic presenting foetuses.
4. Those who gave their consent.

Exclusion Criteria:

1. Co-existing medical illnesses such as diabetes mellitus, cardiac disease, haemoglobinopathies, renal diseases, hypertensive disease, Bronchial asthma,
2. Women currently taking Propranolol or a chronic beta-blocker use
3. Contraindications to labour or vaginal delivery
4. Multiple gestations
5. Preterm labour
6. Chorioamnionitis
7. Known fetal anomalies
8. Abnormal fetal presentation.
9. Antepartum haemorrhage.
10. Contraindication to induction and augmentation of labour
11. Multi-party
12. Known allergy to propranolol

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Induction/Augmentation delivery intervals at delivery | Time frame in minutes from the onset of initiation of Oxytocin to the delivery of the placenta
  Labor acceleration at delivery

SECONDARY OUTCOMES:
Maternal Blood pressure change in mmgh | Change over 30 minutes
  Maternal Blood pressure is checked prior to initiation of oxytocin and 30 minutes after initiation of oxytocin. the difference is noted
Fetal heart rate change in seconds | Change over 30 minutes
  Fetal heart rate is checked prior to initiation of oxytocin and 30 minutes after initiation of oxytocin. the difference is noted

CONTACTS AND LOCATIONS:
Overall Officials: UGOJI DR DARLINGTON-PETER, PART 1, Principal Investigator — ALEX EKWUEME FEDERAL UNIVERSITY TEACHING HOSPITAL, ABAKALIKI, EBONYI STATE, NIGERIA
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
until after defence of the work

REFERENCES:
- [Background] Freedman SB, Adler M, Seshadri R, Powell EC. Oral ondansetron for gastroenteritis in a pediatric emergency department. N Engl J Med. 2006 Apr 20;354(16):1698-705. doi: 10.1056/NEJMoa055119. PMID 16625009